CLINICAL TRIAL: NCT02939911
Title: Residual Neuromuscular Blockade in Paediatric Patients Before Extubation and in Postanesthetic Care Unit:Prospective Observational Cohort Study
Brief Title: Residual Neuromuscular Blockade in Pediatric Anesthesia
Acronym: REPEB
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, doc.MD.Ph.D, Brno University Hospital
Other Study IDs: KDAR FN Brno 2016/2
Record Dates: First submitted 2016-10-18; First posted 2016-10-20 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Residual Neuromuscular Blockade
Keywords: Residual neuromuscular blockade
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Accelerometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Paediatric patients after NMBA administration: Paediatric patients undergoing surgery with neuromuscular blockade
  Interventions: Device: Residual neuromuscular blockade measurement

INTERVENTIONS:
Device: Residual neuromuscular blockade measurement — Just prior extubation in OR and at the arrival to PACU the residual neuromuscular blockade will be measured by accelerometry
  Other Names: accelerometry

SUMMARY:
Residual neuromuscular blockade (RNB) is frequent and it is associated with postoperative morbidity and mortality. The incidence of the RNB in pediatric anesthesia is currently not known. The aim of this prospective observational cohort study is to evaluate the early RNB just before extubation and late RNB at the time of arrival to postanesthetic care unit (PACU).

DETAILED DESCRIPTION:
Residual neuromuscular blockade (RNB) is frequent and it is associated with negative impact on postoperative morbidity and mortality. The incidence of the RNB in adult is well described, however in pediatric subpopulation it is currently not known. The aim of this prospective observational cohort study is to evaluate the early RNB just before extubation and late RNB at the time of arrival to postanesthetic care unit (PACU). In the trial will be enrolled all pediatric patients (28 weeks of age and older - 19 years old) whom will be administered neuromuscular blocking agent during anesthesia. The demographic data will be collected including: age, weight, type of surgery, ASA status. The anesthesia management will be described including: airway management, type and cumulative dose of neuromuscular blocking agent (NMBA) and time and dose of the last administered bolus of NMBA. The residual neuromuscular blockade will be measured according to the standards: TOF Watch accelerometry at the moment prior to extubation (two measurements) in TOF mode and at the arrival to postanesthetic care unit (PACU) (two measurements) in TOF mode.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients undergoing surgery with neuromuscular blocking agents were administered with the age limits

Exclusion Criteria:

* weight under 3000 grams
* neuromuscular disease
* haemodynamic impairment (vasopressor need)
* planned postoperative mechanical ventilation

Ages: 29 Weeks to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Paediatric patients undergoing surgery with neuromuscular blocking agents were administered
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2017-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Early residual neuromuscular blockade | before extubation
  Just prior extubation the residual neuromuscular blockade will be measured by accelerometry

SECONDARY OUTCOMES:
Late neuromuscular blockade | at arrival to PACU
  At the arrival to PACU the residual neuromuscular blockade will be measured by accelerometry

CONTACTS AND LOCATIONS:
Locations (1):
- Brno University Hospital, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Yes